CLINICAL TRIAL: NCT06021847
Title: Effect of Ozone Water in Treatment of Denture Inflammation
Brief Title: Ozonated Water in Treatment of Denture Stomatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Asmaa Nabil Elboraey, Associate Professor of Removable Prosthodontics, National Research Centre, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4447082022
Record Dates: First submitted 2023-08-27; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2022-07

CONDITIONS: Denture Stomatitis
Keywords: Ozonated water; denture stomatitis; Chlorhexidine mouthwash
MeSH Terms: conditions — Stomatitis, Denture

STUDY DESIGN:
Intervention Model Description: Two groups ( complete denture wearers with oral stomatitis). Group I treated with ozonated water while group II treated with chlorhexidine mouthwash.
Who Masked: Participant
Masking Description: The patients didn't know which treatment they received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I patients treated with ozonated water (Active Comparator): The patients were used ozonated water as mouth wash for treatment of denture associated oral stomatitis.
  Interventions: Other: Ozonated water
- Group II patients treated with chlorhexidine mouthwash (Active Comparator): The patients were used chlorhexidine mouth wash for treatment of denture associated oral stomatitis
  Interventions: Other: Chlorhexidine mouthwash

INTERVENTIONS:
Other: Ozonated water — ozonated water was prepared with a concentration of (2-4 mg/l) ozone for 1 min. in a 25 mg of double distilled water 37o C employing an Ozone generator (Ozone generator type N 1888A, China.)
  Arms: Group I patients treated with ozonated water
Other: Chlorhexidine mouthwash — Commercial available chlorhexidine mouthwash in the market was used.
  Arms: Group II patients treated with chlorhexidine mouthwash

SUMMARY:
The effect of Ozonated water on the treatment of oral stomatitis associated with complete denture wearer in comparison to Chlorhexidine mouthwash

DETAILED DESCRIPTION:
Compete denture wearers having oral denture stomatitis were divided into two groups. group I used Ozonated water while group II used Chlorhexidine mouthwash. The growth of Candida albicans, the degree inflammation and pain grade were evaluated before starting the treatment then every week till one month. Also

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous male patients wearing heat cured acrylic resin removable prosthesis.
* Patients having denture associated oral stomatitis.
* Healthy patients free of any systemic diseases.

Exclusion Criteria:

* Smoker patients.
* Patients suffering from any auto immune or systemic diseases, Temporo-mandibular joint disorder ( TMJ disorders and parafunctional oral habits.
* Patients with a history of radiotherapy or chemotherapy.
* Patients having oral lesions.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Candida albicans colonies | day one, 7th day, 14th day and 30th day
  The number of Candida albicans forming units (CFU) was used to assess the effect of two types of treatments.

SECONDARY OUTCOMES:
-Evaluation of inflammation and pain grade | day 1, and 30th day
  - Evaluation of inflammation and pain grade by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa N, Elboraey, Ass,Pro, Principal Investigator — National Research Centre, Egypt
Locations (1):
- National Research Centre, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No